CLINICAL TRIAL: NCT01838252
Title: Hyaluronic Acid Gels for Lower Lid Retraction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Rootman, MD, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-001629
Record Dates: First submitted 2013-04-18; First posted 2013-04-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Ectropion
Keywords: Ectropion; Hyaluronic Acid; Keratoconjunctivitis Sicca; Lower eyelid retraction
MeSH Terms: conditions — Ectropion; Keratoconjunctivitis Sicca | interventions — Hyaluronic Acid; Restylane; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic acid (Experimental): Patients in this arm will receive hyaluronic acid fillers to the lower lid.
  Interventions: Procedure: Hyaluronic acid
- Saline (Sham Comparator)
  Interventions: Procedure: Saline

INTERVENTIONS:
Procedure: Hyaluronic acid — Hyaluronic acid filler will be injected in to the lower lid, elevating it to a more anatomic position
  Other Names: Restylane
  Arms: Hyaluronic acid
Procedure: Saline — Saline will be injected in to the lower lid, elevating it to a more anatomic position
  Arms: Saline

SUMMARY:
Lid retraction is a difficult problem encountered in oculofacial plastic surgery. It can result from previous surgery, radiotherapy or cicatrizing disease or it may be idiopathic. Whatever the aetiology, the cosmetic appearance is troublesome to patients and, can be damaging to the cornea. The definitive therapy for lid retraction is surgical, and often involves complicated procedures including tissue grafting.

Hyaluronic acid gels (HAG) have been FDA approved for the treatment of facial rhytids by subcutaneous injection and volume addition. These gels have gained wide popularity in for cosmetic applications in filling volume deficit areas. Functional applications in the periorbital area have also been described including the filling of volume deficit anophthalmic orbits, ectropion and loagophthalmos. Additionally, pilot studies have found HAG to be useful in correcting both upper and lower eyelid retraction, with good effect.

The purpose of this investigation is to define the clinical utility of HAG correction of lower eyelid retraction in terms of anatomic (lid position), quantitative (dry eye signs on cornea) and qualitative effects (symptom severity).

Our hypothesis is that HAG correction of lower eyelid retraction will improve patient comfort, clinical signs of dry eye and aesthetic self image.

ELIGIBILITY:
Inclusion Criteria:

1. Lower eyelid retraction of >1mm in one or both eyes.
2. Complaints of either significant ocular symptoms (OSDI>13) or cosmetic deformity associated with the eyelid retraction.

Exclusion Criteria:

1. Age less than 21 years: due to lack of data on safety for HAG fillers in pediatric population
2. Age over 65 years of age: as HAG filler effect may be different in this population
3. Are pregnant or nursing: as there is little safety data on potential teratogenicity of HAG fillers
4. Have a demonstrated allergy to HAG fillers or lidocaine
5. Have a current infection, skin sore, pimple, rash, hive or cyst over the injection site: to avoid worsening the infection or transmitting it
6. Have a bleeding disorder or currently taking blood-thinning medications such as Coumadin or heparin on a daily basis.
7. Currently active stage Thyroid Eye Disease

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Lower eyelid position | 6 weeks
  Decrease in inferior scleral show

SECONDARY OUTCOMES:
Subjective dry eye symptoms | 6 weeks
  Ocular surface disease index score
Objective dry eye signs | 6 weeks
  NEI dry eye score
Objective dry eye signs | 6 weeks
  Oxford staining score

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Rootman, MD, MSc, Principal Investigator — University of California, Los Angeles
Locations (1):
- Jules Stein Eye Institute, Los Angeles, California, United States